CLINICAL TRIAL: NCT05277415
Title: Translational and Clinical Aspects of Metabolic, Anabolic and Endothelial Dysfunction in Herat Failure
Brief Title: Translational and Clinical Aspects of Metabolic, Anabolic and Endothelial Dysfunction in Heart Failure
Acronym: MetAnEnd-HF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lars Lund (Other)
Responsible Party: Sponsor-Investigator, Lars Lund, Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008/1:12
Record Dates: First submitted 2022-01-25; First posted 2022-03-14 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction HFrEF
Keywords: cardiac output
MeSH Terms: interventions — Ghrelin

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, parallellel intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ghrelin infusion (Active Comparator): Ghrelin infusion 30 pmol/kg/min, 0.50 ml/min during 120 minutes
  Interventions: Biological: Ghrelin
- Placebo (Placebo Comparator): Saline 0.50 ml/min during 120 minutes
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ghrelin — Ghrelin infusion
  Arms: Ghrelin infusion
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
In patients with HF cardiac output, metabolism and endothelial function will be studied during and after treatment with ghrelin infusion

DETAILED DESCRIPTION:
In patients with HF cardiac output, metabolism and endothelial function will be studied during and after treatment with ghrelin infusion (single dose).

The following parameters will be collected: routine clinical parameters, endothelial function, cardiac structure and function by echocardiography, non-invasively assessed cardiac output and hemodynamics, serologic and of cardiac and renal function, sympathetic and RAS activation, metabolism, anabolic hormone function, inflammation, fibrosis, oxidative stress and apoptosis.

15 patients each group in are adequate to detect a difference between groups and before vs after ghrelin administration in metabolism, anabolic function and endothelial function with a power of 90% and two-sided significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

1. Current or past signs of clinical HF according to the Framingham criteria
2. LVEF<40%
3. NT-proBNP > 300 ng/L

Exclusion Criteria:

1. Inability to or unwillingness to provide informed consent,
2. Participation in research study that involves research drug administration or contraindication to any of the clinically indicated procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Both men and women
Enrollment: 31 (Actual)
Dates: Start 2013-02-17 (Actual); Primary Completion 2014-05-22 (Actual); Study Completion 2014-05-22 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output between treament groups | Procedure (At the end of ghrelin administration)
  Assessed by non-invasive inert gas rebreathing technique (L/min)

SECONDARY OUTCOMES:
Change in endothelial function between treament groups | Procedure (At the end of ghrelin administration)
  Assessed non-invasive by flow mediated dilatory capability of the brachial artery (mm)
Change in cardiac function between treament groups | Procedure (At the end of ghrelin administration)
  Assessed by echocardiography (left ventricular ejection fraction, strain, TAPSE)
GH biomarker | Procedure (At the end of ghrelin administration)
  Circulating biomarkers (GH)
ghrelin biomarker | Procedure (At the end of ghrelin administration)
  Circulating biomarkers ( ghrelin)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lund LH, Hage C, Pironti G, Thorvaldsen T, Ljung-Faxen U, Zabarovskaja S, Shahgaldi K, Webb DL, Hellstrom PM, Andersson DC, Stahlberg M. Acyl ghrelin improves cardiac function in heart failure and increases fractional shortening in cardiomyocytes without calcium mobilization. Eur Heart J. 2023 Jun 9;44(22):2009-2025. doi: 10.1093/eurheartj/ehad100. PMID 36916707